CLINICAL TRIAL: NCT02376751
Title: AN EXPANDED ACCESS PROTOCOL FOR SEBELIPASE ALFA FOR PATIENTS WITH LYSOSOMAL ACID LIPASE DEFICIENCY
Status: No longer available | Type: Expanded Access
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LAL-EA01
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2015-11

CONDITIONS: Lysosomal Acid Lipase Deficiency
Keywords: Cholesteryl Ester Storage Disease; Acid lipase disease; Cholesterol ester hydrolase deficiency; LIPA Deficiency; Wolman disease; Lysosomal Storage Disease
MeSH Terms: conditions — Wolman Disease; Cholesterol Ester Storage Disease; Lysosomal Storage Diseases | interventions — Sebelipase alfa

INTERVENTIONS:
Drug: sebelipase alfa
  Other Names: SBC-102, recombinant human lysosomal acid lipase, rhLAL

SUMMARY:
This is an open-label, multicenter expanded access protocol to allow patients with a confirmed diagnosis of Lysosomal Acid Lipase (LAL) Deficiency in the United States (US), access to sebelipase alfa (recombinant lysosomal acid lipase [rhLAL]) until commercial product is available.

Patients enrolled in the expanded access protocol will receive 1 mg/kg intravenous infusions of sebelipase alfa every other week.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 8 months of age at commencement of treatment with sebelipase alfa.
2. Patient has a confirmed diagnosis of LAL Deficiency.
3. Patient or patient's parent or legal guardian (if applicable) consents to participation in the study. If the patient is of minor age, he/she is willing to provide assent where required per local regulations, and if deemed able to do so.
4. Male and female patients of childbearing potential must use a highly reliable method of birth control (expected failure rate less than 5% per year) from the time they commence treatment through 4 weeks after the last dose of sebelipase alfa.
5. Women of childbearing potential must have a negative serum pregnancy test at commencement of treatment with sebelipase alfa.

Exclusion Criteria:

1. Women who are nursing or pregnant.
2. Patients who received an investigational product within 30 days (for a small molecule) or 60 days (for a biologic) of commencing treatment, and which in the opinion of the investigator or Sponsor, may negatively impact patient safety.
3. Patients who have received sebelipase alfa as part of a clinical trial that is currently active.
4. Patients with known hypersensitivity to eggs.

Min Age: 8 Months | Sex: All
Age Groups: Child, Adult, Older Adult